CLINICAL TRIAL: NCT03548272
Title: POLish Bifurcation Optimal Treatment Strategy (POLBOS 3) Randomized Study
Brief Title: BiOSS LIM C vs 2nd Generation DES in Non-LM Bifurcations
Acronym: POLBOS 3
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Responsible Party: Principal Investigator, Jacek Bil, Principal Investigator, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1.00
Record Dates: First submitted 2018-05-24; First posted 2018-06-07 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Coronary Artery Disease
Keywords: dedicated bifurcation stent; non-LM bifurcation; sirolimus-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BiOSS LIM C (Experimental): Intervention: Percutaneous coronary intervention (PCI) with BiOSS LIM C stent implantation.
  The BiOSS LIM C® is a dedicated bifurcation balloon expandable stent made of cobalt-chromium alloy (strut thickness 70 µm) releasing sirolimus (1.4 µg/mm2) from the surface of a biodegradable coating comprised of a copolymer of lactic and glycolic acids (PGLA). The degradation of the polymer lasts approximately 8 weeks. The BiOSS LIM C® stent consists of two main separate parts with different diameters: wider proximally, and distally smaller. The proximal part is always a bit shorter than the distal one (avg. 1 mm).
  Interventions: Procedure: Percutaneous Coronary Intervention with stent implantation
- regular 2nd generation DES (Active Comparator): Intervention: Percutaneous coronary intervention (PCI) with regular drug-eluting stent implantation (rDES).
  rDES well-tested and available on the market. Xience, Orsiro, Resulte Integrity
  Interventions: Procedure: Percutaneous Coronary Intervention with stent implantation

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention with stent implantation — PCI with BiOSS LIM C or rDES depending on the randomization

SUMMARY:
Coronary bifurcations are encountered in about 15 - 20% of percutaneous coronary interventions (PCI). They are considered technically challenging and associated with worse clinical outcomes than non-bifurcation lesions. Percutaneous coronary intervention (PCI) to the target bifurcation lesion. Randomization (by means envelope randomization) to investigational device: Group 1 for BiOSS LIM C implantation vs Group 2 for any DES implantation.

DETAILED DESCRIPTION:
Single stent implantation in the main vessel-main branch across a side branch is the default strategy (provisional T-stenting, PTS) in all patients enrolled. Bifurcation lesions are assessed according to Medina classification using an index of 1 for stenosis greater than 50% and 0 for no stenosis (visual estimation). There is no restriction regarding lesion length in patient selection. If required, additional stent can be implanted (Alex Plus in the BiOSS Lim C Group). A stent in a side branch (Alex Plus in the BiOSS Lim C Group) should be implanted only if there is proximal residual stenosis greater than 70% after balloon dilatation and/or significant flow impairment after main vessel - main branch stenting and/or a flow limiting dissection.

The implantation protocol for bifurcation is as follows:

1. wiring of both branches;
2. main vessel predilatation and/or side branch predilatation according to the operator's decision;
3. stent implantation (inflation for at least 20 s);
4. proximal optimization technique (POT)
5. side branch postdilatation/side branch stent implantation if necessary
6. final kissing balloon inflation at operator's discretion.
7. Second proximal optimization technique (re-POT)

ELIGIBILITY:
Inclusion Criteria:

1. Subject at least 18 years of age.
2. Subject able to verbally confirm understandings of risks, benefits of receiving PCI for true bifurcation lesions, and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
3. Target main branch lesion(s) located in a native coronary artery with diameter of ≥ 2.5 mm and ≤ 4.5 mm. Target side branch lesion(s) located in a native coronary artery with diameter of ≥ 2.0 mm.
4. Target lesion(s) amenable for PCI with balloon angioplasty of the side branch.

Exclusion Criteria:

1. Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
2. Subjects who refuse to give informed consent.
3. Subjects with LVEF<30%
4. Subjects with moderate or severe degree valvular heart disease or primary cardiomyopathy
5. Distal LM stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Estimated)
Dates: Start 2018-06-12 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
MACE | 12 months
  Major Cardiovascular Events rate (cardiac death, myocardial infarction, target lesion revascularization);

SECONDARY OUTCOMES:
All cause death | 12 months
  All cause death
cardiac death | 12 months
  cardiac death
myocardial infarction | 12 months
  myocardial infarction
target lesion revascularization | 12 months
  target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Invasive Cardiology Central Clinical Hospital of the Ministry of Interior, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Latib A, Colombo A, Sangiorgi GM. Bifurcation stenting: current strategies and new devices. Heart. 2009; 95(6): 495-504. 2. Lassen JF, Holm NR, Stankovic G, et al. Percutaneous coronary intervention for coronary bifurcation disease: consensus from the first 10 years of the European Bifurcation Club meetings. EuroIntervention : journal of EuroPCR in collaboration with the Working Group on Interventional Cardiology of the European Society of Cardiology. 2014; 10(5): 545-560. 3. Collet C, Costa RA, Abizaid A. Dedicated bifurcation analysis: dedicated devices. The international journal of cardiovascular imaging. 2011; 27(2): 181-188. 4. Gil RJ, Vassilev D, Michalek A, et al. Dedicated paclitaxel-eluting bifurcation stent BiOSS(R) (bifurcation optimisation stent system): 12-month results from a prospective registry of consecutive all-comers population. EuroIntervention. 2012; 8(3): 316-324. 5. Bil J, Gil RJ, Vassilev D, et al. Dedicated bifurcation paclitaxel-eluting stent BiOSS Expert(R) in the treatment of distal left main stem stenosis. J Interv Cardiol. 2014; 27(3): 242-251. 6. Vassilev D, Gil R, Milewski K. Bifurcation Optimisation Stent System (BiOSS Lim) with sirolimus elution: results from porcine coronary artery model. EuroIntervention : journal of EuroPCR in collaboration with the Working Group on Interventional Cardiology of the European Society of Cardiology. 2011; 7(5): 614-620. 7. Gil RJ, Bil J, Michalek A, et al. Comparative analysis of lumen enlargement mechanisms achieved with the bifurcation dedicated BiOSS) stent versus classical coronary stent implantations by means of provisional side branch stenting strategy: an intravascular ultrasound study. Int J Cardiovasc Imaging. 2013; 29(8): 1667-1676. 8. Gil R, Bil J, Džavík V, et al. Regular drug-eluting stent versus dedicated coronary bifurcation BiOSS Expert® stent - randomized, multicenter, open-label, controlled POLBOS I trial. Can J Cardiol. 2015; http://dx.doi.org/10.1016/j.cjca.2014.12.024( 9. Gil R, Bil J, Grundeken M, et al. Long-term effectiveness and safety of the sirolimus-eluting BiOSS LIM® dedicated bifurcation stent in the treatment of distal left main stenosis: an international registry. (EuroIntervention - uder review). 2015; 10. Gil RJ, Bil J, Vassiliev D, et al. First-in-man study of dedicated bifurcation sirolimus-eluting stent: 12-month results of BiOSS LIM(R) Registry. J Interv Cardiol. 2015; 28(1): 51-60. 11. Bil J, Gil RJ, Pawlowski T, et al. Assessment of vascular response to BiOSS LIM C(R) stents vs Orsiro(R) stents in the porcine coronary artery model. Cardiovasc Ther. 2017; 12. Medina A, Suarez de Lezo J, Pan M. [A new classification of coronary bifurcation lesions]. Revista espanola de cardiologia. 2006; 59(2): 183. 13. Legutko J, Gil RJ, Buszman P, et al. OCT evaluation of the time course of vessel healing following implantation of new generation biodegradable polymer-coated and sirolimus-eluting cobalt-chromium coronary stent system (ALEX OCT Study). JACC. 2013; 62(18 (S1)): B170-B171. 14. Thygesen K, Alpert JS, Jaffe AS, et al. Third universal definition of myocardial infarction. Circulation. 2012; 126(16): 2020-2035.
- [Derived] Gil RJ, Kern A, Bojko K, Gziut-Rudkowska A, Vassilev D, Bil J. The Randomized, Multicenter, Open-Label, Controlled POLBOS 3 Trial Comparing Regular Drug-Eluting Stents and the Sirolimus-Eluting BiOSS LIM C Dedicated Coronary Bifurcation Stent: Four-Year Results. Biomedicines. 2024 Apr 23;12(5):938. doi: 10.3390/biomedicines12050938. PMID 38790900
- [Derived] Gil RJ, Pawlowski T, Legutko J, Lesiak M, Witkowski A, Gasior M, Kern A, Bil J. Rationale and design of the randomized, multicenter, open-label, controlled POLBOS 3 trial aimed to compare regular drug-eluting stents versus the dedicated coronary bifurcation sirolimus-eluting BiOSS LIM C stent. Medicine (Baltimore). 2019 Apr;98(14):e15106. doi: 10.1097/MD.0000000000015106. PMID 30946377